CLINICAL TRIAL: NCT03651362
Title: Linking Optic Nerve Lesion Length at MRI and the Retinal Axonal Loss at 12 Months From a Clinical Episode of Optic Neuritis
Brief Title: Linking Optic Nerve MRI and the Retinal Axonal Loss After Optic Neuritis
Acronym: IRMANO
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2015_26; 2015-A01159-40 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Optic Neuritis
Keywords: optic neuritis; DIR; visual disability; CIS; multiple sclerosis; NMOSD
MeSH Terms: conditions — Optic Neuritis; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the length of optic nerve lesion on 3D-DIR sequence as an imaging biomarker predictive of retinal axonal loss and visual disability, 12 months after the occurence of a first clinical episode of optic neuritis.

DETAILED DESCRIPTION:
Neurologists and Neuro-Ophthalmologists are in need for reliable and robust imaging biomarkers enabling to predict retinal axonal loss and visual disability after clinical episode of optic neuritis (ON). Length of optic nerve lesion measured on MRI may be one of them.

The aim of our study is to measure the association between the extent of inflammatory demyelinating process on optic nerve at the acute of ON and the retinal degenerative process following optic nerve injury.

The investigators planned to include 50 patients suffering from a recent clinical episode of ON.

Extent of demyelinating inflammatory process will be assessed by the length of optic nerve double inversion recovery (DIR) hypersignal at the acute phase of ON.

The axonal degenerative process following optic nerve demyelinating injury will be assessed by retinal atrophy measured on optical coherence tomography at 12 months after ON, by visual disability measured on low vision contrast acuity scale and by microstructural quality analysis of optic nerve measured on diffusion tensor imaging sequence of the optic nerve.

ELIGIBILITY:
Inclusion Criteria:

* patient suffering from an acute clinical episode of optic neuritis (ON) confirmed by neurophthalmological examination
* < 2 months between start of acute episode of ON and inclusion

Exclusion Criteria:

* past history of homolateral episode of ON
* retinal diseases
* diabeta mellitus
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from a recent clinical episode of ON suggestive of demyelinating disease as clinically isolated syndrome, multiple sclerosis or neuromyelitis optica spectrum disorders.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Severity of retinal axonal loss around papilla after a clinical episode of optic neuritis | 12 months
  peripapillary RNFL thickness decrease

SECONDARY OUTCOMES:
Severity of retinal axonal loss within macula after a clinical episode of optic neuritis | 12 months
  macular volume decrease
Severity of visual disability after a clinical episode of optic neuritis | 12 months
  monocular low contrast (2.5%) vision
Severity of microstructural architecture of optic nerve after a clinical episode of optic neuritis | 12 months
  fractional anisotropy
Progression of optic nerve lesion length | 12 months
  lesion length in mm measured on 3D-double inversion recovery sequence

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Outteryck, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hodel J, Outteryck O, Bocher AL, Zephir H, Lambert O, Benadjaoud MA, Chechin D, Pruvo JP, Vermersch P, Leclerc X. Comparison of 3D double inversion recovery and 2D STIR FLAIR MR sequences for the imaging of optic neuritis: pilot study. Eur Radiol. 2014 Dec;24(12):3069-75. doi: 10.1007/s00330-014-3342-3. Epub 2014 Aug 23. PMID 25149294
- [Background] Miller DH, Newton MR, van der Poel JC, du Boulay EP, Halliday AM, Kendall BE, Johnson G, MacManus DG, Moseley IF, McDonald WI. Magnetic resonance imaging of the optic nerve in optic neuritis. Neurology. 1988 Feb;38(2):175-9. doi: 10.1212/wnl.38.2.175. PMID 3340276
- [Background] Dunker S, Wiegand W. Prognostic value of magnetic resonance imaging in monosymptomatic optic neuritis. Ophthalmology. 1996 Nov;103(11):1768-73. doi: 10.1016/s0161-6420(96)30429-6. PMID 8942868
- [Background] Kallenbach K, Simonsen H, Sander B, Wanscher B, Larsson H, Larsen M, Frederiksen JL. Retinal nerve fiber layer thickness is associated with lesion length in acute optic neuritis. Neurology. 2010 Jan 19;74(3):252-8. doi: 10.1212/WNL.0b013e3181ca0135. PMID 20083802
- [Background] Trip SA, Schlottmann PG, Jones SJ, Altmann DR, Garway-Heath DF, Thompson AJ, Plant GT, Miller DH. Retinal nerve fiber layer axonal loss and visual dysfunction in optic neuritis. Ann Neurol. 2005 Sep;58(3):383-91. doi: 10.1002/ana.20575. PMID 16075460
- [Result] Hadhoum N, Hodel J, Defoort-Dhellemmes S, Duhamel A, Drumez E, Zephir H, Pruvo JP, Leclerc X, Vermersch P, Outteryck O. Length of optic nerve double inversion recovery hypersignal is associated with retinal axonal loss. Mult Scler. 2016 Apr;22(5):649-58. doi: 10.1177/1352458515598021. Epub 2015 Jul 30. PMID 26227005